CLINICAL TRIAL: NCT05654987
Title: Perinatal Mental Health for Refugee Women. An International Study
Brief Title: Perinatal Mental Health for Refugee Women
Acronym: PMH-RW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: University of Gdansk (Other); Taras Shevchenko National University of Kyiv (Other)
Responsible Party: Sponsor
Other Study IDs: 21-PSI-2022
Record Dates: First submitted 2022-11-14; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Perinatal Depression
Keywords: post partum depression; post traumatic stress disorder; anxiety; birth trauma
MeSH Terms: conditions — Depression, Postpartum; Stress Disorders, Post-Traumatic; Anxiety Disorders; Birth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnat women: refugee internal or external pregnant women from Ukraine
- Post partum women: refugee internal or external women during postpartum period (one year after give birth) from Ukranie

SUMMARY:
Since February 24th, 2022, the beginning of Russia's aggression against Ukraine, more than 80,000 women were expected to give birth. Therefore, understanding the impact of war on the perinatal health of women is an important requisite to improve perinatal care.

DETAILED DESCRIPTION:
In general, even in non-war conditions, the perinatal period (from pregnancy to the first year after childbirth) is a vulnerable time. The onset and recurrence of mental disorders are high - it is estimated that 1 in 5 women would develop a perinatal mental disorder with perinatal depression, anxiety disorders, and posttraumatic stress disorder (PTSD) as the leading diagnoses. The experience of war and forced migration may double the risk for mothers and infants. It is highlighted that the experience of war or forced refuge and the associated stress, anxiety, and destabilization have various long-lasting negative consequences for mental health, with high prevalence rates of depression and post-traumatic stress disorder (PTSD). According to clinicians working with the refugee population, a group of pregnant women and new mothers is an especially vulnerable group of the migrant population "in a precarious situation in a foreign country, when the sense of inner homelessness can easily develop, the capacity for empathy and intuitive parenting can be weakened. This may destabilize the maternal/parental function". Studies conducted in war-affected Syria indicated a high percentage (28.2%) of women scoring higher on the postpartum depression scale . Also, according to other studies, high maternal anxiety is associated with a twofold increase in the risk of probable mental disorders in children. The war experience is also a risk factor for adverse, negative pregnancy and childbirth outcomes. It can result in premature birth and low birth weight, which is also observed in a population exposed to armed conflict. However, the rate of preterm births, stillbirths and miscarriages depends on direct exposure to conflict. For example, the adverse outcomes are often related to exposure to chemicals, radiation, exhaust fumes, contaminated water, or food during wartime.

The main aim of this prospective study is to investigate the impact of the war on perinatal mental health: depression, anxiety, post-traumatic stress and birth trauma symptoms on the course of the pregnancy and postpartum period. And also aim to assess the possible protective factors (such as personality traits, social support, sociodemographic characteristics, and access to medical/mental health services ). The research will focus on the two groups of war-affected women in the perinatal period: war refugees in European countries (external refugees) and women who decided to stay in Ukraine (in the same place of residence or as internal refugees).

ELIGIBILITY:
The inclusion criteria at baseline are:

.Being pregnant or a biological mother of a child till twelve months of age or younger.

.Women 18 years of age or older.

.Being a war refugee from Ukraine (entrance to UE countries from 24.02.22) or staying in Ukraine after/during the war.

.Consenting to participate in the study.

The exclusion criteria are:

. Not being currently pregnant or not being the biological mother of a child 12 months of age or younger.

.Women younger than 18 years of age.

. Not consenting to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of women during the perinatal period. The rationale is to evaluate women throughout their pregnancy, and during 1 year after childbirth
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | baseline
  The Edinburgh Postnatal Depression Scale (EPDS) (Cox et al., 1987) This scale includes ten items which assess symptoms of sadness, anxiety and thoughts related to death. The scores range goes from 0 to 30. The cut-off values of 10 or higher and 13 or higher are most often used to identify women who might have depression. 13 has been shown the most useful cut off point established by reviews of international
Generalized anxiety disorder screener GAD- 7 | baseline
  Generalized anxiety disorder screener GAD- 7 (Spitzer, Kroenke, Williams, Löwe, 2006).
  The GAD-7 total score ranges from 0 to 21. The scale's total score indicates the level of anxiety symptoms, with higher scores reflecting a greater anxiety severity. Scores of 5, 10 and 15 represent cut-off points for mild, moderate and severe anxiety, respectivel. When screening for an anxiety disorder, a recommended cut-off point for referral for further evaluation is ten or greater
Impact of Event Stress-Revise | baseline
  A revised version of the Impact of Event Stress-Revised by Weiss and Marmar (1997) The revised version of the Impact of Event Scale (IES-r) has seven additional questions and a scoring range of 0 to 88.
  On this test, scores that exceed 24 can be quite meaningful. 24 or more - PTSD is a clinical concern. Those with scores this high who do not have full PTSD will have partial PTSD or at least some of the symptoms. 33 and above - This represents the best cutoff for a probable diagnosis of PTSD 37 or more
Ten-Item Personality Inventory | baseline
  Ten-Item Personality Inventory ( (Gosling, Rentfrow, and Swann Jr., 2003) The scores range for each scale is from 2 to 14 (two points on each scale; the scores range for each point is from 1 to 7
City Birth Questionnaire | baseline
  City Birth Questionnaire (Ayers et al., 2018) aims to assess PTSD symptoms associated with childbirth according to DSM-5 criteria. It contains 29 items related to the DSM-5 diagnostic criteria, and the remaining two questions are related to the DSM-IV criteria. This questionnaire aims to determine the subjective feeling of discomfort related to a specific traumatic event. The scores range from 0 to 60. AS the authors has pointed out the scores for percentiles are: 25th = 3, 50th = 9, 75th = 18

CONTACTS AND LOCATIONS:
Overall Officials: Maria F. Rodriguez, Professor, Principal Investigator — UNED
Locations (2):
- Magdalena Chrzan-Dętkoś, Gdansk, Poland
- Lyudmyla Krupelnytska, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chrzan-Dętkoś, M., Rodríguez-Muñoz, M. F., Krupelnytska, L., Morozova-Larina, O., Vavilova, A., López, H. G., Murawaska, N., and Radoš, S. N. (2022). Good Practices in Perinatal Mental Health for Women during Wars and Migrations: A Narrative Synthesis from the COST Action Riseup-PPD in the Context of the War in Ukraine. Clínica y Salud, 33(3), 127 - 135. https://doi.org/10.5093/clysa2022a14
- [Derived] Rodriguez-Munoz MF, Chrzan-Detkos M, Uka A, Garcia-Lopez HS, Krupelnytska L, Morozova-Larina O, Vavilova A, Molotokas A, Murawska N, Le HN. The impact of the war in Ukraine on the perinatal period: Perinatal mental health for refugee women (pmh-rw) protocol. Front Psychol. 2023 Mar 13;14:1152478. doi: 10.3389/fpsyg.2023.1152478. eCollection 2023. PMID 36993880